CLINICAL TRIAL: NCT03518424
Title: Scottish Football Injury Study (S-FIS): Epidemiology of Injuries in Scottish Professional Football - A Multi-club, One Season Study
Brief Title: Injury Epidemiology Within Scottish Professional Football
Acronym: S-FIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heriot-Watt University (Other)
Responsible Party: Principal Investigator, Robert McCunn, Performance Sports Manager, Heriot-Watt University
Other Study IDs: S-FIS
Record Dates: First submitted 2018-04-25; First posted 2018-05-08 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Injury;Sports
Keywords: Association football; Soccer; Injury; Epidemiology
MeSH Terms: conditions — Athletic Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present study is to establish the injury incidence, severity and burden typically observed within Scottish professional football clubs. In line with the well-established model of sports injury prevention research proffered by van Mechelen, the first stage in this process is establishing the extent of the problem i.e. injury incidence, severity and burden. Such a multi-club study has never been conducted within Scotland despite a thriving professional game.

ELIGIBILITY:
Inclusion Criteria:

* Professional football player contracted to an SPFL club

Exclusion Criteria:

* Loss of professional status as a footballer

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Scottish Professional Football League (SPFL) club contracted football players
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Injury incidence | 1 year
  The number of injuries per 1000 hours of exposure
Injury type | 1 year
  The types of injuries observed e.g. contact/non-contact, anatomical location, soft-tissue/hard-tissue
Injury burden | 1 year
  The number of days lost due to injury per 1000 hours of exposure

CONTACTS AND LOCATIONS:
Overall Officials: Robert McCunn, Principal Investigator — Oriam: Scotland's Sports Performance Centre
Locations (1):
- Oriam: Scotland's Sports Performance Centre, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.